CLINICAL TRIAL: NCT00148876
Title: A Multicenter Randomized Phase III Study to Compare Capecitabine Alone or in Combination With Trastuzumab in Patients With HER2 Positive Metastatic Breast Cancer and Progression After Previous Treatment With Trastuzumab
Brief Title: TBP Study With Capecitabine Plus Minus Trastuzumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 26; BIG3-05
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer
Keywords: Progression after treatment with Trastuzumab; Metastatic Breast Cancer; Palliative Study
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine (Active Comparator): Capecitabine 2500 mg/m² orally day 1-14 q day 22 until progression and discontinuation of Trastuzumab.
  Interventions: Drug: Capecitabine
- Capecitabine and Trastuzumab (Experimental): Capecitabine 2500 mg/m² orally day 1-14 q day 22 until progression + Trastuzumab 6 mg/kg body weight every 3 weeks i.v. as a 90 min infusion until progression
  Interventions: Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 2500 mg/m² orally day 1-14 q day 22
Drug: Trastuzumab — Trastuzumab 6 mg/kg body weight every 3 weeks i.v.
  Arms: Capecitabine and Trastuzumab

SUMMARY:
This study is done in patients having Breast Cancer with metastasis (patients with positive receptor HER2) whose disease progressed after receiving Trastuzumab.

The primary objective of this study is to compare the time until disease progression between the Treatment Arm CAPECITABINE and the Treatment Arm CAPECITABINE + TRASTUZUMAB

The study has also other secondary and tertiary objectives.

DETAILED DESCRIPTION:
Trial design:

Prospective, multi-center, controlled, non blinded, randomized phase III Study

Treatment:

Patients with HER2 positive metastatic breast cancer and progression after previous treatment with trastuzumab are being randomized to either:

A. Capecitabine 2500 mg/m² orally day 1-14 q day 22 until progression * and discontinuation of Trastuzumab

B. Capecitabine and Trastuzumab:

Capecitabine 2500 mg/m² orally day 1-14 q day 22 until progression * Trastuzumab 6 mg/kg body weight every 3 weeks i.v. as a 90 min infusion until progression *

Objectives:

Primary objective:

To compare the time to disease progression in patients with HER2 positive metastatic breast cancer and progression after previous treatment with trastuzumab randomized to capecitabine alone or in combination with trastuzumab.

Secondary objectives:

To compare the objective response rate between the two arms To compare the duration of response To compare the clinical benefit defined as CR, PR, or stable disease > 24 weeks between the two arms To evaluate the safety of the capecitabine + trastuzumab combination To compare overall survival between the two arms

Tertiary objective:

To determine the HER2 status in tissue collected directly before study entry

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Pathologically confirmed carcinoma of the breast.
3. Locally advanced or metastatic stage of disease not suitable for surgery or radiotherapy alone.
4. HER2-overexpression of the primary or metastatic tumor tissue detected by immunohistochemistry (DAKO) 3+ or gene namplification detected by FISH. HER2-positive primary tumours with HER2-negative metastasis can be included.
5. Disease progression during or after previous chemotherapy and trastuzumab treatment as follows (Trastuzumab has to be given previously for at least 12 weeks, treatment free interval of trastuzumab for a maximum of 6 weeks):

   * Taxanes + trastuzumab given as adjuvant therapy
   * Taxanes + trastuzumab given as first line therapy for palliation
   * Trastuzumab given as first line therapy for palliation alone or in combination with chemotherapeutic agents other than capecitabine or taxanes
6. No more than 1 chemotherapy for palliation (max. Adriamycin dose < or = 400 mg/m²; Epirubicin < or = 600 mg/m²)
7. Patients must have either measurable or nonmeasurable target lesions according to the RECIST criteria (see Appendix 6)
8. At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation portal or there must be pathologic proof of progressive disease
9. At least 4 weeks since major surgery with full recovery.
10. Complete radiology and tumor measurement work up within 4 weeks prior to registration:
11. Karnofsky performance status evaluation > or = 60%
12. Age >18 years.
13. Absolute neutrophil count > or =1,500 cells/microL, platelet count > or =100,000 cells/microL.
14. Bilirubin < or = 2x the upper limit of normal for the institution (ULN); elevation of transaminases and alkaline phosphatase < 2.5x ULN or <5x ULN for patients with liver metastases.
15. Creatinine < or = 2.0 mg/dl.
16. Left ventricular ejection fraction (LVEF) by cardiac ultrasound of > or = 50%.
17. If of childbearing potential, pregnancy test is negative. In addition the patient agrees to use an effective method to avoid pregnancy for the duration of the study.

Exclusion criteria:

1. Known hypersensitivity reaction to the compounds or incorporated substances or known dihydropyrimidine dehydrogenase deficiency.
2. Concurrent immunotherapy or hormonal therapy (antihormonal, contraceptive and/or replacement therapy). Bisphosphonates may be continued.
3. Parenchymal brain metastases, unless adequately controlled by surgery and/or radiotherapy with complete resolution of symptoms and of all steroids.
4. Life expectancy of less than 3 months.
5. Serious intercurrent medical or psychiatric illness that may interfere with the planned treatment (including severe pulmonary conditions, AIDS and serious active infection).
6. History of congestive heart failure or other significant uncontrolled cardiac disease.
7. History of other malignancy within the last 5 years which could affect the diagnosis or assessment of breast cancer.
8. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
9. Treatment with sorivudine or derivates e.g. brivudin
10. Pregnant or nursing women.
11. Male patients.
12. The patient must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre which could be the Principal or Co- investigator's site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2003-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Any progression of disease or disease related death of a patient

SECONDARY OUTCOMES:
Any response documented according to the RECIST Criteria
Time from CR or PR until progression of disease or death due to any cause
Any response and stable disease of >24 weeks duration documented according to the RECIST Criteria
Any grade III/IV toxicity (NCI-CTC version2.0).Premature treatment discontinuation
Any death of a patient

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, Prof. Dr., Principal Investigator — German Breast Group Forschungs GmbH
Locations (1):
- Johann Wolfgang Goethe Universität, Universitätsfrauenklinik, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Click here for more information about this study: TBP Study — http://www.germanbreastgroup.de